CLINICAL TRIAL: NCT00122369
Title: Self Hypnotic Relaxation As An Adjunct To Local Anesthesia During Large Core Breast Biopsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elvira Lang, Former Associate Professor of Radiology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DAMD 17-01-1-0153; 2001P-001681
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer; Anxiety; Pain
Keywords: Breast; Biopsy; Hypnosis; Relaxation; Anxiety; Pain; Medical and Surgical Procedures
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Self-hypnotic Relaxation (Experimental): A research assistant displayed defined behaviors of empathic attention and read to the patient a self-hypnotic relaxation script. Patients also received lidocaine as local anesthetic which is the standard care approach and not considered a unique intervention in terms of the trial.
  Interventions: Behavioral: Self-hypnotic Relaxation; Behavioral: Empathic Attention
- Standard Care (No Intervention): Patients received the routine standard treatment which included application of lidocaine as local anesthetic. This is not considered a unique intervention in terms of the trial. Omitting local anesthetic actually would have been an intervention deviating from routine care.
- Empathic Attention (Active Comparator): A research assistant displayed defined behaviors of empathic attention. Patients also received lidocaine as local anesthetic which is the standard care approach and not considered a unique intervention in terms of the trial.
  Interventions: Behavioral: Empathic Attention

INTERVENTIONS:
Behavioral: Self-hypnotic Relaxation — A research assistant read to the patient a self-hypnotic relaxation script while displaying empathic attention.
  Other Names: Comfort Talk®
  Arms: Self-hypnotic Relaxation
Behavioral: Empathic Attention — A research assistant displayed defined behaviors of empathic attention.
  Other Names: Empathy; Advanced Rapport Skills
  Arms: Empathic Attention; Self-hypnotic Relaxation

SUMMARY:
Percutaneous large core image-guided breast biopsy is a well established tool in diagnosing breast cancer, but the associated anxiety and pain can tax the coping mechanism of even well functioning individuals. Unabated stress during an invasive procedure not only interferes with smooth progression of the ongoing procedure, but can also have deleterious effects when patients need additional procedures and dread recurrent medical traumatization. The long-term objective of this research is to provide patients with a simple coping strategy at the vulnerable time of large core biopsy in the hope that this behavioral intervention will carry over to recovery and future medical procedures. In the largest prospective randomized study of its kind, the researchers showed that a self-hypnotic intervention during percutaneous, image-guided vascular and renal interventions resulted in less pain and anxiety, greater hemodynamic stability, and fewer procedure interruptions. The positive effects of the short initial hypnotic intervention, which was structured in the procedure room, became more pronounced the longer the procedure lasted and carried over into the immediate post-procedure recovery. The investigators therefore challenge the current paradigms that long-lasting effects require intensive presurgical preparation.

DETAILED DESCRIPTION:
Large core image-guided breast biopsy is a well established tool for diagnosing breast cancer. Using ultrasound or X-ray guidance, a large hollow needle is inserted through the skin into the breast and abnormal tissue is removed for diagnosis. Although this procedure is much less invasive than open surgery, it can induce pain and anxiety that can tax the coping mechanism of even the highest functioning individuals. Unrelieved stress during a medical procedure not only interferes with smooth progression of the ongoing procedure, but can also have deleterious effects when patients need additional procedures and feel dread in anticipation. The long-term objective of this research is to provide patients with a simple coping strategy at the time of large core biopsy, when they need it most. The hope is that this newly learned ability to handle distress will carry over to recovery and to future medical procedures. In a prior clinical trial (Lancet 2000:335:1486-1489), the largest prospective randomized study of its kind, the researchers showed that a self-hypnotic intervention during image-guided interventions of the blood vessels and the kidneys resulted in less pain and anxiety, fewer worrisome increases and decreases of blood pressure and heart rate, and fewer procedure interruptions. The positive effects of the short initial hypnotic intervention, which was structured in the procedure room, became more pronounced the longer the procedure lasted and carried over into the immediate post-procedure recovery. Based on these past findings, the researchers therefore predict to show evidence contrary to the current thinking that long-lasting effects require intensive presurgical preparation.

The researchers propose to pursue three interrelated specific aims:

* (Aim 1): Determine the acute effects of self-hypnotic relaxation on pain and anxiety. Strictly defined methods of self-hypnotic relaxation (Group I), will be tested against empathic attention (Group II) and the routine standard of care (Group III) in a prospective randomized study with 240 patients undergoing large core breast biopsy. The impact of the treatment will be validated by comparing during the procedure among groups subjective measures of pain and anxiety as well as objective physiologic indicators of pain and anxiety (frequency of significant increases in heart rate and blood pressure).
* (Aim 2): Determine the delayed effects of self-hypnotic relaxation. Patients' levels of pain, anxiety, and stress will be recorded through days 1-5 after the biopsy and compared among groups. Stress levels measurements will be based on an objective test (the amount of the stress hormone cortisol in the patient's saliva).
* (Aim 3): Determine the effect of the initial self-hypnotic relaxation on distress with upcoming subsequent surgery in women with proven breast cancer. When patients have to return for surgery because their biopsy revealed malignant cells, they will be given questionnaires assessing their degree of perceived stress , anxiety, and preoccupation with their upcoming surgery. Comparison among groups will show the durability of the initial hypnotic intervention.

The researchers hypothesize that:

* Self-hypnotic relaxation reduces pain and anxiety during large core breast biopsy
* Self-hypnotic relaxation at the time of biopsy reduces post-biopsy stress
* Teaching patients coping skills at the critical time of the breast biopsy reduces the patients' distress with upcoming breast surgery.

Upon completion, a short periprocedural self-hypnotic intervention will be validated by rigorous and practical assessment in 240 patients. The relative performance of self-hypnotic relaxation will be known compared to standard care and empathic controls in a well-characterized population of patients with a standardized biopsy wound. The durability of an intervention given at the earliest possible moment of breast cancer diagnosis will be established. This opens the way to future study designs addressing long-term effects on health behavior and psycho-physiologic phenomena.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for large core breast biopsy in the Radiology Department at the Beth Israel Deaconess Medical Center Boston.

Exclusion Criteria:

Patients are excluded if :

* They are unable to give informed consent, or pass screening for impaired mental function or psychosis.
* They are unable to hear or understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2002-03; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira V Lang, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Lang EV, Berbaum KS, Lutgendorf SK. Large-core breast biopsy: abnormal salivary cortisol profiles associated with uncertainty of diagnosis. Radiology. 2009 Mar;250(3):631-7. doi: 10.1148/radiol.2503081087. PMID 19244038
- [Result] Lang EV, Berbaum KS, Faintuch S, Hatsiopoulou O, Halsey N, Li X, Berbaum ML, Laser E, Baum J. Adjunctive self-hypnotic relaxation for outpatient medical procedures: a prospective randomized trial with women undergoing large core breast biopsy. Pain. 2006 Dec 15;126(1-3):155-64. doi: 10.1016/j.pain.2006.06.035. Epub 2006 Sep 7. PMID 16959427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2002 and March 2004, 240 eligible patients were recruited and randomly assigned to treatments. Four patients (including the only male) withdrew after entering the biopsy suite before starting with the intervention in the Intervention Groups or data collection in the Standard Care Group.
Groups:
- Standard of Care: As standard care, the biopsy team attempted to comfort patients in their usual way: they warned of upcoming stimuli, asked patients about their experience, commiserated with them about discomfort, and generally expressed sympathy.
- Empathic Attention: The Empathy condition was defined by a set of structured attentive behaviors engaged in by a research assistant. These behaviors were standardized according to a manual and proven suitable for invasive procedures in radiology (Lang and Berbaum 1997; Lang et al. 1999)
- Self-Hypnotic Relaxation: In the Hypnosis condition, patients received all of the attentive behaviors used in the Empathy condition. In addition, the research assistant read a standardized hypnotic induction script (Lang et al. 1999), and, as needed, addressed the patient's anxiety, pain, or worries according to the prescriptions of the script.
Period: Overall Study
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Started | 76 | 82 | 78
Completed | 76 | 82 | 78
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation | Total
Number analyzed (Participants) | 76 | 82 | 78 | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 69 | 74 | 73 | 216
  >=65 years | 7 | 8 | 5 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.4) | 48.0 (13.22) | 47.8 (13.7) | 48.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 82 | 78 | 236
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 82 | 78 | 236

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety to 10=worst possible anxiety. Patients self-reported anxiety at the beginning (time 0), every 10 minutes, and at the end of their biopsy procedure on a 0-10 numeric verbal anxiety scale (0=no anxiety at all, 10=worst possible anxiety). Participants were followed for the duration of the biopsy procedure, an average of 43 min.
Time Frame: 0 min
Population: Intention to Treat; patients on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 76 | 82 | 78
units on a scale | 4.5 [2 to 6] | 5 [3 to 7] | 5 [3 to 6]

2. Secondary Outcome: Salivary Cortisol Secretion
Description: Secretion of cortisol over time is customarily described in terms of a slope with the time of day of cortisol measurement as the x variable and the natural logarithm of the measured cortisol concentration as the y variable. Cortisol slope is expressed as the natural logarithm of cortisol (micrograms per deciliter) per hour, with 1g/dL corresponding to 27.8 nmol/L. In general, greater negative slopes (with steeper decreases from high morning values to low evening values) are considered better adapted and healthier than flatter (less negative) slopes.
Time Frame: Patients were followed for the 5 days following their breast biopsy
Population: Women learned their diagnosis between Day 1 and 6 (mean day 2.4). Analysis was truncated at day 5 when sufficient numbers of patients for meaningful analysis were available in each group: 16 in the "known malignant" group, 37 in the "known benign" group, and 73 in the "uncertain group" totaling 126 patients.
Measure: Mean (95% Confidence Interval); unit: ln (microgram/dL)/hr
Groups:
- Known Benign Disease: Women who were diagnosed to have benign disease
- Known Malignant Disease: Women who were diagnosed to have malignant disease
- Uncertain Diagnosis: were in the "uncertain" diagnostic group, either because their result had not been communicated yet (n=54); their LCBB could not be performed for technical reasons and they were waiting for a surgical excision (n=14); or histology showed at risk lesions (n=4) or benign cells with surgery recommended for excision and final diagnosis (n=1).
Arm/Group | Known Benign Disease | Known Malignant Disease | Uncertain Diagnosis
Number analyzed (Participants) | 37 | 16 | 73
ln (microgram/dL)/hr | -0.154 [-0.197 to -0.111] | -0.110 [-0.147 to -0.073] | -0.092 [-0.113 to -0.072]
Statistical Analysis 1: Comparison: Known Benign Disease vs Uncertain Diagnosis; The impact of knowing or not knowing the diagnosis became so overwhelming and group composition with regard of whether and which result had been communicated changed daily in the post-biopsy follow-up, so that the originally planned analysis of the impact of Self-Hynotic Relaxation or Empathic Attention on cortisol measures became underpowered. Therefore we focused on the analysis of the impact of diagnosis; Test type: Superiority or Other; p = 0.014, t-test, 2 sided — Bonferoni correction was made so that results with p<0.0167 are considered significant
Statistical Analysis 2: Comparison: Known Malignant Disease vs Uncertain Diagnosis; Test type: Superiority or Other; p = 0.421, t-test, 2 sided — Bonferoni correction was made so that results with p<0.0167 are considered significant
Statistical Analysis 3: Comparison: Known Benign Disease vs Known Malignant Disease; Test type: Superiority or Other; p = 0.138, t-test, 2 sided — Bonferoni correction was made so that results with p<0.0167 are considered significant

3. Secondary Outcome: Impact of Event Scale (IES-15)
Description: The IES is a measure of subjective distress for any specific life event. This 15-item self-report instrument is used to assess experiences of intrusive thoughts (Intrusion subscale) and attempts to consciously avoid such experiences (Avoidance subscale) that are commonly associated with subjective distress about life situations. Answers are given in four ratings from not at all (score 0) to often (score 5), with a possible TOTAL overall range of scores from zero to 75.
  ≥26 indicates moderate to severe distress) of women who at the time of return for breast surgery after their initial biopsy
Time Frame: Patients were followed for up to 3 weeks after their biopsy until the time of their surgery
Population: These 19 patients were the only ones who could be captured for their return to surgery after their initial biopsy.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 7 | 4 | 8
Scores on a Scale | 25 (10.7) | 27 (13.7) | 24 (15)
Statistical Analysis 1: Comparison: Standard of Care vs Empathic Attention vs Self-Hypnotic Relaxation; The null-hypothesis was that there would be no difference among groups; Test type: Superiority or Other; p = 0.56, ANOVA

4. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 10 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 76 | 81 | 77
units on a scale | 4 [2 to 6] | 4 [2 to 7] | 4 [2 to 6]

5. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 20 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 76 | 81 | 75
units on a scale | 4 [2 to 6] | 4 [2 to 7] | 3 [2 to 5]

6. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 30 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 70 | 72 | 66
units on a scale | 4 [2 to 6.5] | 4.5 [2 to 6] | 4 [2 to 6]

7. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 40 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 59 | 57 | 52
units on a scale | 5 [3 to 7] | 5 [3 to 6] | 4 [1.25 to 6]

8. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 50 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 42 | 45 | 39
units on a scale | 6 [2.75 to 7] | 4 [2 to 6] | 3 [1 to 5]

9. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 60 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 32 | 31 | 26
units on a scale | 5 [2.25 to 8] | 4 [2 to 6] | 2.5 [0 to 5.25]

10. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 70 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 23 | 23 | 20
units on a scale | 5 [3 to 8] | 3 [2 to 6] | 2.5 [0 to 4]

11. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 80 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 15 | 12 | 8
units on a scale | 5 [2 to 8] | 4 [2 to 6] | 3 [0 to 4.75]

12. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 90 min
Population: Patients remaining on procedure table (please note that the data in the hypnosis group encompass only 4 patients since the 5th patient did not indicate her anxiety level at that time point)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 8 | 7 | 5
units on a scale | 5 [0.5 to 8.75] | 7 [1 to 8] | 0.5 [0 to 4]

13. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 100 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 7 | 5 | 5
units on a scale | 4 [0 to 9] | 3 [0 to 5.5] | 2 [0 to 5]

14. Primary Outcome: Anxiety Ratings at Specified Time Point During the Procedure
Description: Self-reported anxiety on a scale of 0-10 with 0=no anxiety and 10=worst possible anxiety
Time Frame: 110 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 4 | 2 | 1
units on a scale | 4.5 [0.5 to 8.5] | 2 [0 to 3] | 5 [5 to 5]

15. Primary Outcome: Time Trends of Anxiety Experience
Description: Ordinal regression analysis looks at data as a series of possible splits of patient responses and assesses the odds of experiencing a value at or above as compared to the split; e.g. the probability of experiencing self-reported anxiety scores of 0 vs 1-10; 0-2 vs 3-10 ; 0-4 vs 5-10 etc with anxiety scores reported between 0=no anxiety and 10=worst possible anxiety. The summary analysis with logit slopes gives in the time trend estimate the cumulative probabilities of the response categories over the variable N=procedure time (min). Positive slopes indicate increasing scores above the split point over time, negative slopes indicate decreasing scores, and flat lines no significant change. In the proportional odds model, an encompassing slope - a probability function of linear trend - is generated that not only applies to the logit forms of the individual splits but to the logic forms of graphs that portray all other splits. The resultant slopes then facilitate comparison among groups.
Time Frame: 0-110 min
Population: Intent to Treat; patients undergoing breast biopsy
Measure: Number; unit: logit slopes
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 76 | 82 | 78
logit slopes | 0.18 | -0.04 | -0.27
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority or Other; p < 0.001, Ordinal regression
Statistical Analysis 2: Comparison: Empathic Attention; Test type: Superiority or Other; p = 0.45, Ordinal regression
Statistical Analysis 3: Comparison: Self-Hypnotic Relaxation; Test type: Superiority or Other; p < 0.001, Ordinal regression
Statistical Analysis 4: Comparison: Standard of Care vs Empathic Attention; Test type: Superiority or Other; p < 0.01, Proportional odds model
Statistical Analysis 5: Comparison: Standard of Care vs Self-Hypnotic Relaxation; Test type: Superiority or Other; p < 0.001, Proportional odds model
Statistical Analysis 6: Comparison: Empathic Attention vs Self-Hypnotic Relaxation; Test type: Superiority or Other; p < 0.01, Proportional odds model

16. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 0 min
Population: Intent to Treat; patients on procedure table. (Please note that the data in the empathy group encompass 81 data points since one patient did not indicate her pain level at that time point).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 76 | 82 | 78
units on a scale | 0 [0 to 1.75] | 0 [0 to 0] | 0 [0 to 1]

17. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 10 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 76 | 81 | 77
units on a scale | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 2]

18. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 20 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 76 | 81 | 75
units on a scale | 1 [0 to 4] | 0 [0 to 2] | 0 [0 to 2]

19. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 30 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 70 | 72 | 65
units on a scale | 2 [0 to 4] | 0 [0 to 3] | 0 [0 to 2]

20. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 40 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 59 | 57 | 52
units on a scale | 2 [0 to 5] | 2 [0 to 4] | 0 [0 to 3]

21. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 50 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 41 | 45 | 39
units on a scale | 4 [0 to 6] | 2 [0 to 4.5] | 1 [0 to 3]

22. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 60 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 32 | 31 | 26
units on a scale | 2.5 [0 to 4] | 2 [0 to 5] | 1 [0 to 6]

23. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 70 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 23 | 23 | 20
units on a scale | 4 [2 to 6] | 2 [0 to 4] | 2 [0 to 4.5]

24. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 80 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 15 | 12 | 8
units on a scale | 5 [2 to 7] | 3.5 [1.25 to 4.75] | 2.5 [0 to 7]

25. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 90 min
Population: Patients remaining on procedure table. (Please note that the data in the hypnosis group encompass 4 data points since one patient did not indicate her anxiety level at that time point).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 8 | 7 | 5
units on a scale | 5 [5 to 8] | 2 [1 to 5] | 1.5 [0 to 7.5]

26. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 100 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 7 | 5 | 5
units on a scale | 9 [7 to 9] | 2 [1 to 4.5] | 2 [0.5 to 5.5]

27. Primary Outcome: Pain Ratings at Specified Time Point During the Procedure
Description: Self-reported pain on a scale of 0-10 with 0=no pain at all and 10=worst possible pain
Time Frame: 110 min
Population: Patients remaining on procedure table
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 4 | 2 | 1
units on a scale | 8.5 [8 to 9.75] | 3 [3 to 3] | 10 [10 to 10]

28. Primary Outcome: Time Trends of Pain Experience
Description: Ordinal regression analysis looks at data as a series of possible splits of patient responses and assesses the odds of experiencing a value at or above as compared to the split; e.g. the probability of experiencing self-reported pain scores of 0 vs 1-10; 0-2 vs 3-10 ; 0-4 vs 5-10 etc with pain scores reported between 0=no pain, and 10=worst possible pain. The summary analysis with logit slopes gives in the time trend estimate the cumulative probabilities of the response categories over the variable N=procedure time (min). Positive slopes indicate increasing scores above the split point over time, negative slopes indicate decreasing scores, and flat lines no significant change. In the proportional odds model, an encompassing slope - a probability function of linear trend - is generated that not only applies to the logit forms of the individual splits but to the logic forms of graphs that portray all other splits. The resultant slopes then facilitate comparison among groups.
Time Frame: 0-110 min
Population: Intent to Treat; patients undergoing breast biopsy
Measure: Number; unit: logit slopes
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Number analyzed (Participants) | 76 | 82 | 78
logit slopes | 0.53 | 0.37 | 0.34
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority or Other; p < 0.001, Ordinal regression
Statistical Analysis 2: Comparison: Empathic Attention; Test type: Superiority or Other; p < 0.001, Ordinal regression
Statistical Analysis 3: Comparison: Self-Hypnotic Relaxation; Test type: Superiority or Other; p < 0.001, Ordinal regression
Statistical Analysis 4: Comparison: Standard of Care vs Empathic Attention; Test type: Superiority or Other; p = 0.024, Proportional odds model
Statistical Analysis 5: Comparison: Standard of Care vs Self-Hypnotic Relaxation; Test type: Superiority or Other; p = 0.018, Proportional odds model
Statistical Analysis 6: Comparison: Empathic Attention vs Self-Hypnotic Relaxation; Test type: Superiority or Other; p = 0.73, Proportional odds model

ADVERSE EVENTS:
Time Frame: Patients were followed for up to one week after their biopsy
Description: Adverse event reporting was done using the Reporting Standard of the Society of Interventional Radiology
Arm/Group | Standard of Care | Empathic Attention | Self-Hypnotic Relaxation
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/82 | 0/78
Other Adverse Events (participants affected / at risk) | 7/76 | 11/82 | 3/78
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=76) | Empathic Attention (N=82) | Self-Hypnotic Relaxation (N=78)
Hematoma (Surgical and medical procedures) | 5 (5) | 9 (9) | 3 (3)
Vasovagal episode (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
For the assessment of the Secondary Outcome parameter we were able to recruit only 19 women whom we could contact early enough on the day of their breast cancer surgery to fill out the IES. This limits the power of the statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No